CLINICAL TRIAL: NCT05590936
Title: Comparison of the Effectiveness of Dimenydrinate vs Ondasetron on the Prevention of Postoperative Nausea and Vomiting
Brief Title: Dimenydrinate vs Ondansetron for PONV (DONV)
Acronym: DONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 52699
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: PONV in Laparoscopic Cholocystectomies
MeSH Terms: interventions — Dimenhydrinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dimenydrinate (Active Comparator): Preoperative per os administration of 50 mg dimenydrinate
  Interventions: Drug: Dimenhydrinate Tablets
- Ondasentron (Other): Intraoperative intravenous administration of 4 mg ondansetron
  Interventions: Drug: Ondansetron iv

INTERVENTIONS:
Drug: Dimenhydrinate Tablets — 2 hours preoperative per os administration of 50 mg dimenhydrinate
  Arms: Dimenydrinate
Drug: Ondansetron iv — Intraoperative intravenous administration of 4 mg ondansetron
  Arms: Ondasentron

SUMMARY:
This study will investigate the impact of dimenydrinate (H1-receptor antagonist) versus ondansetron (HT3-receptor antagonist) in postoperative nausea and vomiting, in surgery-related preoperative stress and in the incidence of postoperative complications that could lengthen the LOS in PACU and/or the overall LOS.

DETAILED DESCRIPTION:
Dimenydrinate has been extensively used for motion sickness. However, as far as postoperative nausea and vomiting is concerned the results are still conflicting.

This study will investigate the impact of dimenydrinate (H1-receptor antagonist) versus ondansetron (HT3-receptor antagonist) in postoperative nausea and vomiting, in surgery-related preoperative stress and in the incidence of postoperative complications that could lengthen the LOS in PACU and/or the overall LOS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* ASA PS I-III
* Undergoing laparoscopic general surgery operations or laparoscopic gynecological operations

Exclusion Criteria:

* Refused to participate
* Age other than 18-75 years old
* Pregnant patients
* Non-elective operations
* Patients that are not able to receive p.os agents
* Medical history of Brugada Sdr or Brugada-like/related ECG abnormalities
* Long-Qt Sdr or concurrent use of medications that may cause long-QT ECG abnormalities
* Medical or family history of psychosis
* Allergy in dimenydrinate or in dimenydrinate drug versions
* Perioperative use of dexamethasone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
PONV | 30 minutes postoperative
  PONV recording in patients undergone laparoscopic cholocystectomy
PONV | 60 minutes postoperative
  PONV recording in patients undergone laparoscopic cholocystectomy
PONV | 12 hours postoperative
  PONV recording in patients undergone laparoscopic cholocystectomy
PONV | 24 hours postoperative
  PONV recording in patients undergone laparoscopic cholocystectomy

SECONDARY OUTCOMES:
preoperative anxiety | 24 hours before operation
  preoperative anxiety recording in patients undergone laparoscopic cholocystectomy measured by one hundred points scale
preoperative anxiety | 30 minutes before operation
  preoperative anxiety recording in patients undergone laparoscopic cholocystectomy measured by one hundred points scale
Awaken time | on extubation
  time from anesthetic drug cessation until extubation

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly; Konstantinos George Stamoulis, MD, PhD, Study Director — University Hospital of Larissa
Locations (1):
- University Hospital of Larisa, Department of Anesthesiology, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided